CLINICAL TRIAL: NCT04903964
Title: The Effect of Individualized Nutrition Training Given to the Families of Children With Congenital Heart Disease (CHD) in the Post-Operative Period on Their Growth and Development
Brief Title: Growth and Development of Children With Congenital Heart Disease (CHD)
Acronym: CHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Emel Yürük, Lecturer, Cukurova University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: Adana Cukurova University
Record Dates: First submitted 2021-04-30; First posted 2021-05-27 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Researcher-Subject Relations
Keywords: Child Health and Nursing; Congenital Heart Disease; Family Centered Care; Growth and Development; İndividual Nutrition Education.
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Intervention Model Description: The research is a randomized controlled experimental study.
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- oral nutrition only group that received nutrition education (Experimental): This group consists of children who are fed orally according to their chronological age. The questionnaire form developed by the researcher and the parameters used in the evaluation of growth (height, head and chest circumference measurement) and Ankara Development Screening Inventory (AGTE) will be applied to the child and his / her family included in the specified group. Nutrition education prepared by the researcher will be given to the mothers of the children included in this group. After the nutrition training given to their mothers, the growth and development monitoring parameters of the child, body weight, height, head and chest circumference, will be repeated at regular intervals. Ankara Development Screening Inventory (AGTE) will be applied. The follow-up frequency of the hospitalized child after the operation will be determined and the measurements will be checked.
  Interventions: Other: family-centered nutrition education
- group that received nutrition education and fed with nutritional support (Experimental): This group consists of children who receive nutritional support provided by oral food supplements, oral food supplements, enteral tube feeding and / or parenteral nutrition. The questionnaire form developed by the researcher and the parameters used in the evaluation of growth (height, head and chest circumference measurement) and Ankara Development Screening Inventory (AGTE) will be applied to the child and his / her family included in the specified group. Nutrition education prepared by the researcher will be given to the mothers of the children included in this group. After the nutrition training given to their mothers, the growth and development monitoring parameters of the child, body weight, height, head and chest circumference, will be repeated at regular intervals. Ankara Development Screening Inventory (AGTE) will be applied. The follow-up frequency of the child hospitalized after the operation will be determined and the measurements will be checked.
  Interventions: Other: family-centered nutrition education
- control group (No Intervention): While collecting research data on the specified dates; Comparison group (KG) will be selected as many as the number of volunteers who want to participate in the research. No nutritional attempt will be made to the child included in this group. The parameters used in the evaluation of growth (height, head and chest circumference measurement) and the Ankara Development Screening Inventory (AGTE) will be applied to children aged 0-3 who are followed up due to congenital heart disease.

INTERVENTIONS:
Other: family-centered nutrition education — There is a training program prepared by the researcher to increase the nutritional knowledge of mothers with children aged 0-3. The definition and importance of nutrition in the session, respectively, adequate and balanced nutrition, insufficient and unbalanced nutrition damages, grouping of nutrients, feeding 0--6 months old baby, feeding premature baby, breastfeeding, situations to be considered while breastfeeding, starting additional foods, 9-12 monthly baby nutrition, 1-3 years old child nutrition and nutritional nutrition support.
  Arms: group that received nutrition education and fed with nutritional support; oral nutrition only group that received nutrition education

SUMMARY:
The Effect of Individualized Nutrition Training Given to the Families of Children with Congenital Heart Disease (CHD) in the Post-Operative Period on their Growth and Development This study was conducted experimentally to determine the effects of individualized nutrition training given to mothers of children who had surgery for CHD on their growth and development.

DETAILED DESCRIPTION:
The Effect of Individualized Nutrition Training Given to the Families of Children with Congenital Heart Disease (CHD) in the Post-Operative Period on their Growth and Development This study was conducted experimentally to determine the effects of individualized nutrition training given to mothers of children who had surgery for CHD on their growth and development.

The data of the study were collected at Çukurova University Medical Faculty Balcalı Hospital Cardiovascular Surgery between 20/01/2021-30/06/2021. The research was conducted by interviewing the families of 42 children with congenital heart disease. Personal information form, growth parameters and Ankara Developmental Screening Inventory were applied to three groups formed as two experimental and control groups by randomization method. Family-centered care and individualized nutrition training were applied to the first experimental group who was fed orally and and the second experimental group orally and nutritionally fed. These trainings were about nutritional contents suitable for the age of the baby, the way of preparing the food and meeting the calorie needs of the baby. No training was given to the control group during the research process. The growth and development parameters of all three groups were evaluated and the effect of education was examined.

ELIGIBILITY:
Inclusion criteria:

* Congenital heart disease,
* Born on time (38-42 weeks)
* Over 2.300 gr.
* fed with additional nutritional support to oral and oral nutrition,
* Decided to have surgery,
* 0-3 years old,
* The children and their families who were followed up in the post-operative service were included.

Exclusion criteria:

* No congenital heart disease
* Not planned to have surgery,
* over 3 years old,
* Children with additional congenital malformation, dysmorphic syndrome, chromosomal disease, severe infection, hypothyroidism and similar disorders that may cause growth and development retardation were excluded from the study.

Ages: 30 Days to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Body weight measurement of growth parameter | every weeek up to 1 months
  In order to determine the physical growth status of the babies, kilograms (in kg) will be measured by the researcher. These measurement results will be given as average Z scores ((kg) type and percentile values. Body weight is measured on an Oncomed electronic scale by removing the clothing and subtracting the dry weight of the ultra-prima brand diaper.

SECONDARY OUTCOMES:
Height measurement of growth parameter | every weeek up to 1 months
  Height (in cm) will be measured by the researcher to determine the physical growth status of the babies. These measurement results will be given as average Z-scores (cm) type and percentile values. For height measurement, a head-foot board (infantometer) with a measuring tape is used.
Head circumference measurement of growth parameters | every weeek up to 1 months
  The head circumference (in cm) will be measured by the researcher to determine the physical growth state of the babies. These measurement results will be given as average Z scores (cm) type and percentile values. Head circumference measurement is made with an inelastic tape measure from the most protruding point of the occipital bone over the ear and over the line passing over the eyebrows.

CONTACTS AND LOCATIONS:
Overall Officials: EMEL YÜRÜK, Principal Investigator — ÇUKUROVA ÜNİVERİSTESİ
Locations (1):
- Çukurova Üniversitesi Balcalı Hastanesi, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
planned to be completed as a thesis
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: When the thesis research is finished, it will be used for publication as an article publication
Access Criteria: 2 year
URL: https://www.cbs.dk/en/research/cbs-research-profile/research-data-management/research-data-management-plans